CLINICAL TRIAL: NCT03310632
Title: A Phase I/II Study to Determine the MTD and to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of Antroquinonol in Combination With SOC in First Line Metastatic Pancreatic Cancer
Brief Title: Determine Function of Antroquinonol in Combination With SOC in First Line Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHPanc-1-001
Record Dates: First submitted 2017-10-01; First posted 2017-10-16 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Neoplasm
Keywords: Antroquinonol; Hocena; metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — antroquinonol

STUDY DESIGN:
Intervention Model Description: Phase I
  Run-in DDI and dose escalation:
  Six patients will be enrolled in the run-in DDI cohort of the dose-escalation part of the study (ie, Cohort 1) and 3 to 6 patients may be enrolled in Cohort 2. The total number of patients to be entered in the dose-escalation part of this study will depend on the emergence of DLTs at each dose level, but will be up to 12 if no replacement occurs at the 2 predefined dose levels.
  Phase II
  Cohort expansion:
  Up to an additional 40 patients may be enrolled at the MTD or MFD/RD. A power calculation was not employed to determine the sample size of the study, as this is aproof of concept study with a preliminary assessment of anti-tumor activity of antroquinonol in combination with nab-paclitaxel + gemcitabine in metastatic pancreatic cancer patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antroquinonol with SOC (Experimental): Antroquinonol will first be conducted by dose escalation(200mg TID and 300mgTID) to characterize the safety of antroquinonol in combination with the standard of care (SOC) (nab-paclitaxel + gemcitabine) and to identify the MTD of antroquinonol in patients with metastatic pancreatic cancer.
  At the cohort expansion part of the study, up to an additional 40 patients will be enrolled at the MTD or MFD/RD.
  Interventions: Drug: Antroquinonol

INTERVENTIONS:
Drug: Antroquinonol — Antroquinonol: 100 mg and corn oil 100 mg encapsulated in a gelatin capsule administered orally. Dose will be selected(200mg TID or 300mg TID with SOC) after phase I, then follow up the best dose for 40 Patients for the efficacy.
  Other Names: Hocena

SUMMARY:
Antroquinonol is proposed for the treatment of neoplasms. The proposed clinical trial is a Phase I/II study designed to evaluate antroquinonol in combination with nab-paclitaxel and gemcitabine in first line treatment naïve subjects with Stage IV metastatic pancreatic carcinoma. The first part of study will focus on the treatment of pancreatic cancer with 200 mg TID and 300 mg TID, clinical treatment duration of 4 weeks, to determine the MTD or MFD (based on PK and capsules strength) of antroquinonol in combination with a standard dose regimen of nab-paclitaxel and gemcitabine. The extended Phase II will focus on the efficacy of antroquinonol with SOC. Safety and pharmacokinetic profiles will be studied in the proposed clinical trial.

DETAILED DESCRIPTION:
Golden Biotech are planning a Phase I/II study to determine the maximum tolerable dose (MTD) and to evaluate safety/tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of antroquinonol in combination with nab-paclitaxel-gemcitabine in first line metastatic pancreatic cancer.

Phase I

Run-in DDI and dose escalation:

The dose escalation part of the study will be conducted to characterize the safety of antroquinonol in combination with the standard of care (SOC) (nab-paclitaxel + gemcitabine) and to identify the MTD of antroquinonol in patients with metastatic pancreatic cancer. The MTD is the dose level at which <33% (2/6) of patients experience a DLT. Within the dose escalation part of the study, a total of 6 patients will be enrolled in a run-in DDI portion to assess the effect of antroquinonol (a cytochrome P450 [CYP]3A4/CYP2C8 inhibitor) on the PK of paclitaxel (a CYP3A4/CYP2C8 substrate). Patients within this cohort (Cohort 1) will receive treatment as follows:

* Cycle 0 (28-day cycle): nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 (as per SOC) via intravenous (IV) infusion on Days 1, 8, and 15.
* Cycle 1 (28-day cycle): antroquinonol 200 mg administered TID on Days 1 through 28 and nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 via IV infusion on Days 1, 8, and 15.

Intense PK sampling to assess the PK of paclitaxel will be conducted in Cycles 0 and 1. The primary PK endpoints will include Cmax, AUC0-t, and AUCinf. Available bioanalytical data will be assessed in an ongoing manner to assess the effect of antroquinonol on the systemic exposure (Cmax and AUCs) of paclitaxel. Data will be reviewed by the Safety Monitoring Committee (SMC) prior to enrollment of additional patients into the dose-escalation part of the study.

For Cohort 1, the occurrence of DLTs will be assessed from Day 1 to Day 28 of Cycle 1. If ≤1 patient experiences a DLT, dosing in the dose escalation part will proceed. If ≥2 patients experience a DLT, dosing in the dose escalation part of the study will be discontinued. If ≤1 patient in Cohort 1 experiences a DLT then dosing in Cohort 2 of the dose escalation part will proceed as follows: - All Cycles: antroquinonol 300 mg administered TID on Days 1 through 28 and nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 via IV infusion on Days 1, 8, and 15 (ie, 1 cycle = weekly for 3 weeks, then 1 week off) .

Three patients will be enrolled initially into Cohort 2, these patients will be assessed for DLTs within the first 28-day dosing cycle. This cohort will be expanded to 6 total patients if 1 DLT is observed in the first 3 patients within Cohort 2. If ≤1 DLT is observed at the 300 mg dose then the 300 mg dose will be considered the MFD. If >1 DLT is observed at the 300 mg group then 200 mg will be considered the MTD and/or the SMC will review the available data and determine the MTD/recommended dose (RD).

Patients enrolled into the dose escalation part of the study (Cohorts 1 and 2) will continue to receive treatment with antroquinonol (200 or 300 mg, respectively) in combination with nab-paclitaxel + gemcitabine in 28-day cycles at the discretion of the Investigator without a maximum duration until unacceptable toxicity or progressive disease (PD).

The total number of patients to be entered in the dose escalation part of the study will depend on the emergence of DLTs at each dose level and the total number of dose levels investigated. Up to 12 patients are planned to be treated in the dose-escalation part if no patient needs to be replaced for DLT and safety evaluation.

Phase II

Cohort expansion:

During the cohort expansion part of the study, up to an additional 40 patients will be enrolled at the MTD or MFD/RD. The dose level in the cohort expansion phase will not exceed the MTD, or highest safe dose tested in the dose-escalation phase if MTD is not reached. Patients in the cohort expansion will receive treatment as follows:

- All Cycles: antroquinonol at the MTD or MFD/RD administered TID on Days 1 through 28 and nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 via IV infusion on Days 1, 8, and 15 (ie, 1 cycle = weekly for 3 weeks, then 1 week off) .

Patients enrolled into the cohort expansion part of the study will continue to receive treatment with antroquinonol at the MTD or MFD/RD in combination with nab-paclitaxel + gemcitabine in 28-day cycles at the discretion of the Investigator without a maximum duration until unacceptable toxicity or PD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years of age.
2. Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas, measurable according to the RECIST 1.1.
3. Diagnosed with metastatic disease within 6 weeks before enrollment.
4. Treatment-naïve patients with metastatic pancreatic adenocarcinoma who have received no previous systemic therapy (except adjuvant or neoadjuvant therapy if progression occurred >6 months from last treatment or surgery, respectively, and no prior nab-paclitaxel).
5. Adequate hematologic, hepatic, and renal function, including:

   * Hemoglobin ≥9 g/dL
   * Absolute neutrophil count ≥1500/mm3
   * Platelet count ≥100 000/mm3
   * Total bilirubin ≤1.25 × upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤5 × ULN
   * Albumin ≥3 mg/dL
   * Serum creatinine ≤1.5 mg/dL or calculated creatinine clearance ≥50 mL/min as determined by the Cockcroft-Gault equation.
6. ECOG performance status of 0 or 1.
7. For women of childbearing potential, a negative serum pregnancy test result at Screening.
8. Willing to use 2 medically accepted and effective methods of contraception from the list below during the study (both men and women as appropriate) and for 3 months after the last dose of study drug:

   1. Established use of oral, injected, or implanted hormonal methods of contraception
   2. Placement of an intrauterine device or intrauterine system
   3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
   4. Male sterilization (with the appropriate postvasectomy documentation of the absence of sperm in the ejaculate)
   5. True abstinence (when this is in line with the preferred and usual lifestyle of the patient).
9. Patient must be able to provide written informed consent for participation in the study.
10. Life expectancy ≥12 weeks as assessed by the Investigator.

Exclusion Criteria:

1. Islet-cell neoplasms or locally advanced disease.
2. Chemo-, hormone-, or immunotherapy or investigational drug at Screening or prior to enrollment.
3. Treatment with any drug(s) known to be a strong inhibitor or inducer of CYP2C19,CYP3A4, CYP2C8, and CYP2E1 within 14 days of the date of first administration of study drug and during study treatment.
4. Other malignancies diagnosed within the past 5 years (other than curatively treated cervical cancer in situ, nonmelanoma skin cancer, superficial bladder tumors Ta [noninvasive tumor] and TIS [carcinoma in situ], or nonmetastatic prostate cancer Stage 1 to 2, which has been previously treated with surgery or radiation therapy, and serum prostate-specific antigen is within normal limits [test performed within the past 12 months prior to the date of first administration of study drug]).
5. Patients with any serious active infection (ie, requiring an IV antibiotic, antifungal, or antiviral agent).
6. Patients with known human immunodeficiency virus, active hepatitis B, or active hepatitis C.
7. Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the Investigator, would either compromise patient safety or interfere with the evaluation of the safety of the study drug.
8. Known or suspected substance abuse or alcohol abuse.
9. Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs from study treatment, or compromise the ability of the patient to give written informed consent.
10. Inability to swallow oral medications or a recent acute gastrointestinal disorder with diarrhea, (eg, Crohn's disease), malabsorption, or CTCAE Grade >2 diarrhea of any etiology at baseline.
11. Female patients who are pregnant or breastfeeding, or male or female patients of reproductive potential who are not employing an effective method of contraception.
12. Any known hypersensitivity to any component of nab-paclitaxel, gemcitabine, or antroquinonol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD( phase I) | 4 weeks
  The MTD is the dose at which <33% of patients experience a dose limiting toxicity (DLT) within the first 28-day cycle of antroquinonol and nab-paclitaxel
  + gemcitabine combined treatment
tumor assessment in millimeters | 6 months
  measure tumor size by CT or MRI

SECONDARY OUTCOMES:
Body Surface Area in meter^2 | up to 48 weeks
  measure patient's weight and height and calculated by {[Height (cm) × Adjusted Body Weight] × 1/3,600}^1/2
Maximum Plasma Concentration | 3 weeks
  maximum observed plasma concentration of antroquinonol and paclitaxel
Area Under the Curve | 3 weeks
  Plasma concentrations of antroquinonol and paclitaxel will be measured and PK parameters calculated where applicable.
CA19-9 level in units per milli-liter | up to 48 weeks
  blood will be draw and measured. Other emerging antroquinonol biomarkers may be evaluated.
Eastern Cooperative Oncology Group (ECOG) status | up to 48 weeks
  Medical Doctors judged the patient's performance status

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Florida Hospital Tampa, Tampa, Florida
  - CTCA Southeastern Regional Medical Center, Newnan, Georgia
  - Henry Ford Health System, Detroit, Michigan
  - Cancer Treatment Centers of America - Eastern Regional Medical Center, Philadelphia, Pennsylvania
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No